CLINICAL TRIAL: NCT01522261
Title: The Use of Mechanical Bowel Preparation in Pelvic Reconstructive Surgery (MBP)
Brief Title: The Surgical Benefit and Pt.Tolerability Between Two Different Bowel Cleansing Regimens Performed Prior to Pelvic Reconstructive Surgery. Does One Bowel Cleansing Regimen Improve the Surgeons Visual Field Significantly Better Than the Other.
Acronym: MBP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Urogynecology Associates (Other)
Responsible Party: Principal Investigator, Lekha S. Hota, Principal Investigator, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BUA 007-2011
Record Dates: First submitted 2012-01-09; First posted 2012-01-31 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Mechanical Bowel Prep
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mechanical Bowel Prep (Active Comparator): Patients randomized to complete a Mechanical Bowel Prep. (complete bowel cleansing) and fleet enemas prior to surgery.
  Interventions: Other: Mechanical Bowel Prep
- No Mechanical Bowel Prep. (Active Comparator): Patients randomized to complete two fleets enemas only prior to surgery.
  Interventions: Other: No Mechanical Bowel Prep

INTERVENTIONS:
Other: Mechanical Bowel Prep — Patients randomized to MBP will complete procedure per standard instructions.
  Arms: Mechanical Bowel Prep
Other: No Mechanical Bowel Prep — Patient randomized to fleets enemas only prior to surgery
  Arms: No Mechanical Bowel Prep.

SUMMARY:
Does mechanical bowel preparation (complete bowel cleansing)help the Surgeon with visualization of the operative field during laparoscopic pelvic reconstructive surgery?

DETAILED DESCRIPTION:
Patients will be randomized to receive a complete MBP or not prior to their surgical procedure. All patients will use 1 fleets enema the night before surgery and one the morning of surgery to ensure that the rectum is empty of all stool. This will be done since some surgeons use a rectal probe in the rectum to help with manipulation during the procedure. Stool in the rectal vault could contaminate the surgical field and lead to an infection.

Patients will be randomized at their pre-op visit and provided instructions according to the group assignment. On the day of surgery patients will be asked to complete a questionnaire in the pre-op holding area to assess their overnight symptoms including insomnia, weakness, abdominal distention, nausea, thirst and overall tolerability of the Bowel Preparation assigned.

Immediately after surgery, the primary surgeon will be asked to complete a visual analog score sheet evaluating the ease of the procedure with regard to retraction of the large and small bowel to help with visualization of the sacral promontory, retraction from posterior cul-de-sac, and maintaining adequate positioning after retraction. All surgeons (attendings, fellows, and residents) will be blinded re: the patients group assignment. Each primary surgeon will be asked to assign a final grade to the procedure as easy, medium, or difficult based on overall bowel retraction.

At their 2 week follow up visit patients will be asked to report return of bowel function (first bowel movement or flatus) in # of days after surgery and incidents of stool leakage post op.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing the following laparoscopic pelvic reconstructive procedures for pelvic organ prolapse:

* Laparoscopic sacrocervicopexy
* Laparoscopic sacrocolpopexy
* Laparoscopic sacrohysteropexy
* Laparoscopic uterosacral ligament suspension

Who understand and are willing to comply with the study requirements, including agreeing to answer the preoperative and postoperative questionnaires

Exclusion Criteria:

* Previous abdominal or laparoscopic colon surgery (not including transrectal procedures)
* History of abdominal malignancy
* History of surgical debulking for previous malignancy
* Non-english speaking
* Pregnancy
* Hx of abdomino-pelvic radiation
* Contraindications to Sodium Phosphate
* Contraindications to laparoscopic surgery

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
To determine whether there is there an added benefit in using a MBP with regard to positioning of the large and small bowel for exposure of key anatomic structures during pelvic reconstructive surgical procedures. | Surgeons will be asked to complete a questionnaire re: their impressions of the visual field on immediately Post op.
  The primary objective of this protocol is to determine whether there is truly an advantage for the surgeon (visually) in having patients complete a Mechanical Bowel Prep prior to surgery or if an enema completed the evening before and morning of the surgery is sufficient.

SECONDARY OUTCOMES:
To evaluate whether MBP (total bowel cleansing) delays the return of bowel function and/or increases the risk of perioperative leakage of stool (fecal incontinence)post operatively. | We will be following the subject from the day of surgery through 2 weeks post op.

CONTACTS AND LOCATIONS:
Overall Officials: Lekha Hota, M.D., Principal Investigator — Boston Urogynecology Associates
Locations (1):
- Boston Urogynecology Associates, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Adelowo AO, Hacker MR, Modest AM, Apostolis CA, Disciullo AJ, Hanaway KJ, Elkadry EE, Rosenblatt PL, Rogers KJ, Hota LS. The Use of Mechanical Bowel Preparation in Pelvic Reconstructive Surgery: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2017 Jan/Feb;23(1):1-7. doi: 10.1097/SPV.0000000000000346. PMID 27782976